CLINICAL TRIAL: NCT06893978
Title: Placental Organoids Development: Application in the Study of the Human Reproduction Pathophysiology.
Acronym: PLORG
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7203
Record Dates: First submitted 2024-11-20; First posted 2025-03-25 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-11

CONDITIONS: Preeclampsia; Pregnancy Loss; Preterm Birth; Healthy
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Placenta organoids treatment — Placenta organoids in vitro treatment with heparin, aspirin, IVIG, filgrastim and metformin

SUMMARY:
Placental organoids represent an in vitro 3D reconstruction model of the human placenta and of its complex cellular organization to evaluate the pharmacological effect in terms of placentation, gene expression, protein synthesis and placental secretomics.

DETAILED DESCRIPTION:
Placental organoids represent an in vitro 3D reconstruction model of the human placenta and of its complex cellular organization. Placental organoid model can be used in the study of placental pathophysiology. In in particular, it provides a personalized model for sartorial in vitro evaluation of personalized therapeutic efficacy of different pharmacological therapies. In particular, with placental organoid it is possible to evaluate the pharmacological effect in terms of placentation, gene expression, protein synthesis and placental secretomics.

ELIGIBILITY:
Inclusion Criteria:

* Women with uncomplicated normal term pregnancy undergoing elective cesarean section for previous uterine surgery or breech presentation of the fetus;
* Patients with retained abortion and history of recurrent abortion sine causa at the end of the work-up of investigations performed according to ESHRE guidelines, undergoing revision of the uterine cavity;
* Patients diagnosed with preeclampsia, defined in accordance with the definitions of ISSHP, undergoing cesarean section;
* Patients with preterm onset, before 37 weeks gestational age, of spontaneous labor, undergoing cesarean section in labor for low weight or abnormal fetal presentation.

Exclusion Criteria:

* Age <18 years;
* Chronic infection with HIV or HCV;
* Ongoing malignant neoplasms;
* Multiple pregnancies;
* Inability to provide informed informed consent.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with normal pregnancy (n=5) or complicated by:
  * miscarriage (n=5);
  * preeclampsia (n=5);
  * preterm delivery (n=5); afferent to the U.O.C. of Obstetrics of the Agostino Policlinico Universitario Agostino Gemelli IRCCS of Rome.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Development of placental 3D organoid model | From the date of caesarean section until the development of placental organoids, assessed up to 36 months.
  Morphological characteristics of placental 3D organoids successfully developed from placentas obtained from full-term physiological pregnancies and pathological conditions (abortion, preeclampsia, preterm delivery).
  Assessment Parameters: Organoid formation efficiency (%)
Characterization of placental 3D organoid model | From the date of caesarean section until the development of placental organoids, assessed up to 36 months.
  Assessment of cell viability (live/dead staining)
Viability of Placental Organoids | From date of caesarean section until the development of placental organoids, until 36 months
  Measurement of cell proliferation rate in normal and pathological placental organoids before and after anticoagulant, anti-inflammatory, and immunomodulatory treatments (heparin, aspirin, metformin, IVIg, filgrastim).
  Assessment Parameters: Cell viability (live/dead staining)

SECONDARY OUTCOMES:
Gene Expression in Placental Organoids | From date of caesarean section until the development of placental organoids, until 36 months
  Quantification of tissue-specific gene expression in normal and pathological placental organoids before and after treatments.
  Assessment Parameters: Differential expression of target genes (qPCR)
Secretome Analysis of Placental Organoids | From date of caesarean section until the development of placental organoids, until 36 months
  Analysis of extracellular vesicles and soluble factors secreted by placental organoids before and after treatments.
  Assessment Parameters: Quantification of cytokines by ELISA assay
Proliferative Capacity of Placental Organoids | From date of caesarean section until the development of placental organoids, until 36 months
  Assessment of percentage of proliferating cells
Growth capacity of placental organoids | From date of caesarean section until the development of placental organoids, until 36 months
  Assessment of organoid growth rate (diameter increase over time).
Protein expression in placental organoids | From date of caesarean section until the development of placental organoids, until 36 months
  Assessment of differential expression of proteins by Western blot, immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Tersigni, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Ostetricia e Patologia Ostetrica, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No